CLINICAL TRIAL: NCT02740686
Title: Changes in Inflammatory Markers During Pulmonary Rehabilitation Based on Exacerbation States in COPD
Acronym: CIMPRES-COPD
Status: Completed | Type: Observational
Sponsor: University of Lincoln (Other)
Collaborators: National Health Service, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Alex Jenkins, Mr Alex Jenkins, University of Lincoln
Other Study IDs: 16/LO/0865
Record Dates: First submitted 2016-04-08; First posted 2016-04-15 (Estimated); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Exercise; Immunity; Inflammation; Biomarkers
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity; Inflammation | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood samples will be used on the day of collection and analysed before being appropriately disposed of on the same day. Blood samples will be centrifuged with separated plasma to be frozen at -80c for later analysis of cellular content. Sputum samples will also be centrifuged with supernatant extracted and frozen -80c for later analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Frequent exacerbators: Exacerbations will be defined as "a respiratory event which led to a hospitalisation or the prescription of antibiotics and/or oral corticosteroids". Clinicians will ask patients to retrospectively recall how many exacerbations they have had in the past 12 months. Patients will be allocated to the frequent exacerbators group based on whether they have had 2 or more hospitalisations for exacerbations or have taken 2 or more courses on steroids/antibiotics within the past 12 months. Blood sample collection at the following pulmonary rehabilitation sessions: 1st (pre-exercise), 2nd (pre and post-exercise), 8th (pre-exercise), last session (pre and post exercise). Sputum samples collected pre-exercise at the following pulmonary rehabilitation sessions: 1st, 8th, and last session.
  Interventions: Other: Sample collection
- Infrequent exacerbators: Exacerbations will be defined as "a respiratory event which led to a hospitalisation or the prescription of antibiotics and/or oral corticosteroids". Clinicians will ask patients to retrospectively recall how many exacerbations they have had in the past 12 months. Patients will be allocated to the infrequent exacerbators group based on whether they have had no more than 1 hospitalisation for exacerbations or have not taken more than 1 course of steroids/antibiotics within the past 12 months. Blood sample collection at the following pulmonary rehabilitation sessions: 1st (pre-exercise), 2nd (pre and post-exercise), 8th (pre-exercise), last session (pre and post exercise). Sputum samples collected pre-exercise at the following pulmonary rehabilitation sessions: 1st, 8th, and last session.
  Interventions: Other: Sample collection
- Healthy smokers: Recruited in accordance with inclusion/exclusion criteria with no medical history of COPD diagnosis and currently smoke.This group will be recruited by a nurse using medical records to assess smoking status and age-matching to the COPD groups. A resting blood sample will be taken from these patients and used to compare baseline measurements with the COPD groups.
  Interventions: Other: Sample collection
- Healthy never smokers: Recruited in accordance with inclusion/exclusion criteria with no medical history of COPD diagnosis and have never smoked.This group will be recruited by a nurse using medical records to assess smoking status and age-matching to the COPD groups. Resting blood samples will be taken from these patients and used to compare baseline measurements with the COPD groups.
  Interventions: Other: Sample collection

INTERVENTIONS:
Other: Sample collection — Frequent exacerbators and infrequent exacerbators will have blood and sputum samples obtained around pulmonary rehabilitation. No other intervention will be administered. Healthy controls will have resting blood samples taken.

SUMMARY:
This study will examine the inflammatory response to exercise encompassed as part of a standard pulmonary rehabilitation programme in patients with chronic obstructive pulmonary disease (COPD). Patients will be split into two groups, frequent exacerbators or infrequent exacerbators, dependent upon exacerbation history to compare responses to pulmonary rehabilitation amongst phenotypes.

DETAILED DESCRIPTION:
Pulmonary rehabilitation has been proven to benefit COPD patients in terms of quality of life and functional capabilities. The effects of pulmonary rehabilitation (exercise) on immune function are unclear despite clear benefits of exercise on immune function in healthy individuals being identified. Moderate-intensity and frequency of exercise has been shown to decrease the risk of upper respiratory tract infections in healthy individuals in comparison to sedentary individuals. Respiratory infections, also known as exacerbations, in COPD are the main cause of hospitalisation and mortality. Therefore, if exercise can modulate immune function in COPD, it can be encouraged further in COPD to reduce hospitalisation risk. However, it is important to compare the effects of exercise amongst different phenotypes as frequent exacerbators are known to have elevated inflammatory markers, and may consequently respond to exercise differently to infrequent exacerbators, paving a rationale for a different approach to this subset of patients.

ELIGIBILITY:
Inclusion Criteria:

* 58 frequent exacerbators and 58 infrequent exacerbators (116 in total) who have been diagnosed with any severity of COPD (according to BTS criteria, i.e. >10 pack year smoking history and post bronchodilator spirometry FEV1/FVC ratio <0.70 and FEV<80%).

Exclusion Criteria:

* Inability or unwillingness to sign informed consent
* Any unstable ongoing cardiovascular events which may be exacerbated by exercise
* Inability to complete walk tests due to physical or mental impairment
* Other active inflammatory conditions e.g. rheumatoid arthritis, cancer.
* Known asthma, allergic rhinitis or other respiratory disease (bronchiectasis, pulmonary fibrosis)

Healthy control group - Patients who have not been diagnosed with COPD or any other respiratory condition and are characteristically (age (between 45-85 years old) & smoking status) matched to recruited COPD patients.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 116 COPD patients, confirmed by diagnosis, will be recruited (58 frequent and 58 infrequent exacerbators in accordance with criteria listed above) to the study who have been referred to, and are about to enrol, on pulmonary rehabilitation.
  20 healthy smokers and 20 healthy never smokers will be recruited for baseline measurements to compare with COPD patients.
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2016-07; Primary Completion 2018-08-28 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
Concentration of inflammatory markers in plasma and sputum (C-reactive protein, Fibrinogen, Interleukin(IL)-6, IL-8 | July 2016 - August 2018

SECONDARY OUTCOMES:
Changes in the expression of anti-inflammatory genes | July 2016 - August 2018
Total and differential blood leukocyte count | July 2016 - August 2018
Pre-activation and activation of blood neutrophils using flow cytometry | July 2016 - August 2018
Pro-coagulant and pro-inflammatory microparticle signatures in plasma | July 2016 - August 2018
Severe, moderate and mild exacerbations (number of /days to defined events, severity, recovery) | July 2016 - August 2018
Respiratory Symptoms™ (RS-Total score; RS-Breathlessness; RS-Cough and Sputum, and RS-Chest Symptoms) | July 2016 - August 2018
Routine clinical outcome measures following pulmonary rehabilitation (completion rates and clinically important differences - ISWT, ESWT, 6MWD, CRQ) | July 2016 - August 2018
Differences in basal levels of inflammation between frequent and infrequent exacerbators in comparison to healthy controls | July 2016 - August 2018

CONTACTS AND LOCATIONS:
Overall Officials: Alex R Jenkins, MPhil, Principal Investigator — PhD student
Locations (6):
- United Kingdom (6):
  - Lindum Medical Practice, Lincoln, Lincolnshire
  - Nettleham Medical Practice, Lincoln, Lincolnshire
  - Welton Surgery, Lincoln, Lincolnshire
  - Birchwood Medical Practice, Lincoln, Lincolnshire
  - Sudbrooke Drive Community Centre, Lincoln
  - Bracebridge Community Centre, Lincoln

IPD SHARING:
Plan to Share IPD: No